CLINICAL TRIAL: NCT04968236
Title: Application of the Deep Versus Superficial Dry Needling and Stretching Technique in the Treatment of the Quadriceps Rectus Femoris Muscle.
Brief Title: Dry Needling Versus Conservative Treatment in the Rectus Femoris Muscle Approach.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06/2014
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Dry Needling; Stretch; Rectus Femoris Muscle
Keywords: Deep Dry needling; Superficial dry needling; muscle stretching; rectus femoris
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deep dry needling (Experimental): With the subject lying supine, we will first locate a latent myofascial trigger point in the rectus femoris muscle.Subsequently, we will apply a deep dry needling technique to the latent trigger point and make 10-12 incisions.
  Interventions: Other: Deep Dry Needling
- Superficial dry needling (Experimental): With the subject lying supine, we will first locate a latent myofascial trigger point in the rectus femoris muscle.Subsequently, we will apply a superficial dry needling technique to the latent trigger point. Once the needle is placed in the subcutaneous cellular tissue, we manipulate the needle by twisting it until an unpleasant response is provoked. We keep the needle for 5 minutes
  Interventions: Other: Superficial Dry Needling
- Passive muscle stretching (Experimental): With the patient positioned in the supine position, the pelvis stabilized with a strap and the lower extremity where we are going to apply the rectus femoris muscle stretch placed outside the table, we perform a passive stretching technique, increasing hip extension and knee flexion until the patient feels the tension. The position is held for 60 seconds.
  Interventions: Other: passive stretching

INTERVENTIONS:
Other: Deep Dry Needling — In-and-out into different directions technique to encounter sensitive spots in an MTrP region.
  Arms: Deep dry needling
Other: Superficial Dry Needling — This technique involves inserting a needle at a depth that is into the subcutaneous tissue and may be combined with manipulation of the needle while in situ.
  Arms: Superficial dry needling
Other: passive stretching — Type of stretching in which you stay in one position for a set time. In this case, hip extension and knee flexion.
  Arms: Passive muscle stretching

SUMMARY:
In recent years, dry needling techniques have become widespread in the field of musculoskeletal pain treatment. Specifically, the management of myofascial trigger points has been the focus of these techniques.

One of the objectives has been to improve the flexibility of those muscles that, due to the presence of myofascial trigger points, had a decrease in this parameter.

This study aims to determine whether the application of a dry needling technique is more effective than analytical stretching of the muscle.

DETAILED DESCRIPTION:
Hypothesis of the study Deep dry needling of latent trigger points of the rectus femoris produces greater effects on flexibility, strength and pain than superficial dry needling or stretching.

- Overall objective: To compare the differences that occur in flexibility, strength and pain threshold to pressure after the application of deep dry needling, superficial dry needling and stretching on latent trigger points of the rectus femoris.

- Specific objectives To determine the changes produced by deep dry needling on flexibility, strength and pain threshold to pressure.

To determine the changes produced by superficial dry needling on flexibility, strength and pain threshold to pressure.

To determine the changes in flexibility, strength and pain threshold to pressure produced by conventional assisted stretching.

To check if the changes remain after 7 days of the application of the techniques.

To assess the inter-rater reliability of the Goniometer APP in the study sample.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 18 and 65 years old.
2. To have at least 70º of knee flexion.
3. Be aware of and accept the study criteria (informed consent).
4. Healthy subjects, without previous hip or knee pathology or involved musculature.

Exclusion Criteria:

1. To have pain.
2. Having pain in the quadriceps or hip at the time of the study.
3. Currently following physiotherapy or analgesic treatment.
4. Belenophobia (fear of needles).
5. Recent surgery or trauma in the area.
6. Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Knee joint range | Change from baseline at 7 days
  Knee flexion motion assessment by using the Goniometer APP, which is a digital goniometer that has proven its reliability and validity.The overall concordance coefficient has shown very good to excellent with active measurements (range, 0.60-0.97).
Muscle strength | Change from baseline at 7 days
  Force will be measured by a manual dynamometer (microFET®2, Hoggan Scientific LLC). Measurements will be taken in Newtons (N). It will be evaluated in the movements of flexion of knee. Manual dynamometry has proven to be a tool with excellent intra-examiner reliability to assess isometric force in flexion of the knee, with an intraclass correlation coefficient (ICC) of 0.96 (0.93-0.98).

SECONDARY OUTCOMES:
Pressure Pain Threshold (PPT) | Change from baseline at 7 days
  An algometer Wagner FPI 10-WA will be used to determine the PPT in rectus femoris trigger points

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Centro Investigación Fisioterapia y Dolor, Alcalá de Henares, Madrid
  - Physiotherapy and Pain Institute, Alcalá de Henares, Madrid

IPD SHARING:
Plan to Share IPD: No